CLINICAL TRIAL: NCT01382004
Title: Single-dose Azithromycin Versus Penicillin G Benzathine for the Treatment of Yaws in Children
Brief Title: Single-dose Azithromycin for the Treatment of Yaws
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lihir Medical Centre (Other)
Collaborators: Centre For International Health (Other)
Responsible Party: Principal Investigator, Oriol Mitja, M.D., Lihir Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YAWS-AZ01
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Yaws; Treponema Infection; Neglected Tropical Disease
Keywords: Neglected diseases; Children
MeSH Terms: conditions — Yaws; Treponemal Infections; Neglected Diseases | interventions — Penicillin G; Azithromycin; Penicillin G Benzathine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Penicillin-G-Benzathine (Active Comparator): penicillin-G-Benzathine : 50,000 UI/Kg single dose(maximum 2.4 million units IM)
  Interventions: Drug: Penicillin-G-benzathine
- Azithromycin (Experimental): Azithromycin: 30 mg/kg single dose (Maximum: 2.000 mg.)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Penicillin-G-benzathine — Screening examination: Medical history (emphasis on skin lesions and bone signs) Physical examination.Blood samples for VDRL and TPHA. Clinical safety. Laboratory evaluations: haemoglobin, total WBC count, differential WBC count, platelet count, ALT, AST, urea and creatinine.
  Routine assessments: General clinical assessment and physical examination on Days 0 (treatment administered) and 14. Adverse events and concomitant medications (at baseline, Day 14 and in any unscheduled visit). Photograph documentation of skin lesions (at 14 days follow up visit). Follow-up visits performed on 3 and 6 will have a ± 14 days allowable window
  Other Names: Zithromax; Bicillin LA
  Arms: Penicillin-G-Benzathine
Drug: Azithromycin — Screening examination: Medical history (emphasis on skin lesions and bone signs) Physical examination.Blood samples for VDRL and TPHA. Clinical safety. Laboratory evaluations: haemoglobin, total WBC count, differential WBC count, platelet count, ALT, AST, urea and creatinine.
  Routine assessments: General clinical assessment and physical examination on Days 0 (treatment administered) and 14. Adverse events and concomitant medications (at baseline, Day 14 and in any unscheduled visit). Photograph documentation of skin lesions (at 14 days follow up visit). Follow-up visits performed on 3 and 6 will have a ± 14 days allowable window
  Arms: Azithromycin

SUMMARY:
Yaws, an endemic treponematosis and as such a neglected tropical disease (NTD), is currently making a comeback in children in rural areas. Injectable long acting penicillin remains the drug of choice for the treatment of yaws. However, on the basis of successful experience with venereal syphilis in large-scale studies, oral azithromycin has emerged as a potential alternative that overcomes the major medical and logistic disadvantages of the current regimen.

In this non-inferiority randomized clinical trial the investigators propose a comparable scheme for the treatment of yaws, to test the efficacy of a single, oral dose of azithromycin versus a single, i.m. dose of benzathine penicillin G.Sample size has been calculated to detect a non-inferiority margin of 10%. Children < 15 years of age with a confirmed diagnosis of yaws will be randomly assigned to receive 30mg/Kg (maximum 2g) of azithromycin orally or 50.000units/Kg (maximum 2.4MU) of penicillin-G-benzathine intramuscularly. The primary outcome is treatment efficacy, with cure defined serologically (a decline in the VDRL titer of at least two dilutions by six months after treatment) and, in primary yaws, also by epithelialization of ulcers within two weeks.

DETAILED DESCRIPTION:
Regulatory status: Investigational - Randomized Clinical Trial. Registered product for antibacterial therapy

BACKGROUND Penicillin remains the drug of choice for the treatment of endemic treponematoses including yaws. This type of treatment is effective and cheap. There are, however, some disadvantages: the pain associated with a large volume (4 ml) deep i.m. injection, a high prevalence of self-reported allergy to penicillin, structural and logistic problems related to a treatment based on injection of drugs.

Azithromycin, a macrolide antibiotic with a long (68 hours) half-life in tissue and proven efficacy against T.pallidum is a promising candidate. In two randomized trials, for the treatment of syphilis in adults, a single 2-g oral dose of azithromycin achieved cure rates equivalent to that of standard treatment with 2.4 MU of penicillin G benzathine. On the basis of experience with venereal syphilis, azithromycin has emerged as an alternative treatment for Yaws. It represents a more accessible treatment as it could be prescribed by village health workers and therefore enable yaws control to be more easily incorporated into other primary health-care programmes.

The product is available as an oral tablet to be administered at a single dose of 30mg/Kg in children and 2 g in adults. Safety and efficacy using azithromycin 30 mg/kg given as a single dose in the treatment of pediatric patients over 6 months of age with otitis media have been established and approved by the FDA.

INFORMED CONSENT All participants (or their guardian or parents) who are eligible for enrolment in the trial according to biological and demographic inclusion criteria are provided with detailed information on the purpose of the trial and on risks and benefits of participation, according to information listed in an information sheet. Consent is provided in writing.

SAMPLE SIZE JUSTIFICATION

The sample size would be 244; It was calculated on the basis of a non-inferiority trial design and the following assumptions:

Statistical power of 80 percent;to exclude the possibility that the absolute efficacy of azithromycin was at least 10% percent less than that of penicillin; 5% significance level using a one-sided equivalence test of proportions; assuming that the true efficacy of each agent was equivalent at 95 percent and that approximately 10 percent of participants would be lost to follow-up.

RANDOMIZATION PROCEDURE A random allocation schedule, stratified according to study group, will be generated centrally with the use of blocked randomization, random permuted blocks of four, and a 1:1 allocation ratio. The allocation will be concealed from investigators through the use of sequentially numbered, sealed envelopes

ELIGIBILITY:
Inclusion Criteria:

* All children 6 months to 15 years of age who present to LMC with suggestive skin lesions or joint pains and VDRL and TPHA testing are positive
* Suggestive skin lesions defined as: Symptomatic > 4 weeks, painless, a traumatic ulcers with raised margins. VDRL positive when titer of at least 1:16

Exclusion Criteria:

* Pregnancy
* Less than 6 months of age
* Known allergy to penicillin or macrolide
* Use of antibiotics active against treponema during the preceding six months (penicillin-G-benzathine, ceftriaxone, azithromycin or doxycycline)

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Serologic cure | 6 months follow up
  Serologic cure, defined as a decrease in the VDRL titer by at least two dilutions at six month follow-up examination, with the titer at the time of treatment used as the baseline.
  In the case of primary skin lesions, complete resolution or improvement of lesions within two weeks after treatment is also required.

SECONDARY OUTCOMES:
clinical cure | 6 months
  Clinical cure (improvement 14 days after treatment, assessed by photograph comparison over the time)
3 months cure rate | 3 months
  Serological Cure rates three months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Quique Bassat, MD, PhD, Study Director — Centre for International Health Research/Hospital Clínic/University of barcelona
Locations (1):
- Lihir Medical Centre, Kavieng, New Ireland Province, Papua New Guinea

REFERENCES:
- [Derived] Mitja O, Hays R, Ipai A, Penias M, Paru R, Fagaho D, de Lazzari E, Bassat Q. Single-dose azithromycin versus benzathine benzylpenicillin for treatment of yaws in children in Papua New Guinea: an open-label, non-inferiority, randomised trial. Lancet. 2012 Jan 28;379(9813):342-7. doi: 10.1016/S0140-6736(11)61624-3. Epub 2012 Jan 11. PMID 22240407